CLINICAL TRIAL: NCT02943616
Title: ABSORB Post-Approval Clinical Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Abbott has decided to stop selling the Absorb stent which was the product under evaluation in this study.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-307
Record Dates: First submitted 2016-10-19; First posted 2016-10-25 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Ischemic Heart Disease
Keywords: Absorb GT1 BVS; BVS; Bioabsorbable; Myocardial ischemia; Stent thrombosis; Stents
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Absorb BVS (Experimental): Subjects receiving Absorb GT1 Bioresorbable Vascular Scaffold (BVS).
  Interventions: Device: Absorb BVS

INTERVENTIONS:
Device: Absorb BVS — Commercially approved Absorb GT1 BVS, herein referred to as "Absorb".
  * Scaffold diameters: 2.5, 3.0, and 3.5 mm
  * Scaffold lengths: 8, 12, 18, 23 and 28 mm
  Absorb is a temporary scaffold that will fully resorb over time and is indicated for improving coronary luminal diameter in patients with ischemic heart disease due to de novo native coronary artery lesions (length ≤ 24 mm) with a reference vessel diameter of ≥ 2.5 mm and ≤ 3.75 mm.

SUMMARY:
The ABSORB Post-Approval Clinical Study is a prospective, open-label, multi-center, single-arm, non-randomized trial to evaluate the safety of the use of ABSORB in a real-world setting following commercial physician training'and to observe the effectiveness of commercial physician training on appropriate vessel sizing.

DETAILED DESCRIPTION:
After approval of commercial use of Absorb GT1 Bioresorbable Vascular Scaffold (BVS) System in over 75 countries as of December 31, 2015, Abbott Vascular has developed a post-approval commitment plan that includes the initiation of the ABSORB Post-Approval Clinical Study, a single-arm trial that will include approximately 2000 subjects at approximately 265 sites in the US and Canada.

The objectives of ABSORB PostApproval Study are the following:

* Evaluate the safety of the use of Absorb in a real world setting following commercial physician training.
* Observe the effectiveness of commercial physician training on appropriate vessel sizing in the use of Absorb in a real world setting.

The study design allows evaluating low frequency events, effectiveness of commercial physician training and education for very small vessels (< 2.25 mm as assessed by quantitative coronary angiography [QCA]), and confirmation of generalizability of the treatment with Absorb to real-world practice. The estimated follow-up of safety and effectiveness will be 3 years.

Angiographic Subgroup:

Approximately the first 500 consecutive subjects implanted by operators inexperienced in the usage of Absorb GT1 BVS to receive baseline assessment of reference vessel diameter (RVD) by the angiographic core laboratory. An inexperienced operator is defined as having performed two or fewer Absorb implants prior to commercial approval. The purpose of the angiographic subgroup is to evaluate the effectiveness of training in the selection of appropriately sized coronary arteries for GT1 BVS implantation. Study staff will be notified after the procedure if the subject is in the angiographic subgroup, and instructed to send pre-procedure angiogram and supporting materials to core laboratory for assessment.

ELIGIBILITY:
Inclusion Criteria:

* The subject agrees and signs the Institutional Review Board (IRB) approved informed consent form
* The subject receives an Absorb

Exclusion Criteria:

* Subject is a member of a vulnerable population.

Vulnerable population: Defined as subject whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate. Examples of populations which may contain vulnerable subjects include: Individuals with lack of or loss of autonomy due to immaturity or through mental disability, persons in nursing homes, children, impoverished persons, subjects in emergency situations, ethnic minority groups, homeless persons, nomads, refugees, and those incapable of giving informed consent. Other vulnerable subjects include, for example, members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the sponsor, members of the armed forces, and persons kept in detention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiac death, myocardial infarction (CD/MI) | 1 year
  Myocardial infarction will be assessed per the Universal MI definition.

SECONDARY OUTCOMES:
Definite/probable scaffold thrombosis (ST) | 1 year
  ST is assessed per the Academic Research Consortium (ARC) definite/probable definition.
The annual rate of definite/probable scaffold thrombosis | At 1 year post-index procedure
  ST is assessed per the Academic Research Consortium (ARC) definite/probable definition.
The annual rate of definite/probable scaffold thrombosis | Between 1 year and 2 years (366 to 730 days) post index procedure
  ST is assessed per the Academic Research Consortium (ARC) definite/probable definition.
The annual rate of definite/probable scaffold thrombosis | Between 2 years and 3 years (731 to 1095 days) post index procedure
  ST is assessed per the Academic Research Consortium (ARC) definite/probable definition.
Percentage of very small vessels (per-lesion basis) | Pre-procedure (on day 0)
  This is the commercial Training Assessment Endpoint (Angiographic Subgroup only). Pre-procedure reference vessel diameter (RVD) < 2.25 mm as assessed by core laboratory using quantitative coronary angiography (QCA).
Death (Cardiac, Non-Cardiac) | ≤ 7 days post index procedure (In-hospital )
  Cardiac death (CD): Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Death (Cardiac, Non-Cardiac) | 30 days
Death (Cardiac, Non-Cardiac) | 180 days
Death (Cardiac, Non-Cardiac) | 1 year
Death (Cardiac, Non-Cardiac) | 2 years
Death (Cardiac, Non-Cardiac) | 3 years
All Myocardial Infarction (All MI) | ≤ 7 days post index procedure (In-hospital )
All Myocardial Infarction (All MI) | 30 days
All Myocardial Infarction (All MI) | 180 days
All Myocardial Infarction (All MI) | 1 year
All Myocardial Infarction (All MI) | 2 years
All Myocardial Infarction (All MI) | 3 years
Target Lesion Revascularization (TLR) | ≤ 7 days post index procedure (In-hospital )
  TLR is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.
Target Lesion Revascularization (TLR) | 30 days
Target Lesion Revascularization (TLR) | 180 days
Target Lesion Revascularization (TLR) | 1 year
Target Lesion Revascularization (TLR) | 2 years
Target Lesion Revascularization (TLR) | 3 years
Ischemia Driven TLR (ID-TLR) | ≤ 7 days post index procedure (In-hospital )
  TLR is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.
Ischemia Driven TLR (ID-TLR) | 30 days
Ischemia Driven TLR (ID-TLR) | 180 days
Ischemia Driven TLR (ID-TLR) | 1 year
Ischemia Driven TLR (ID-TLR) | 2 years
Ischemia Driven TLR (ID-TLR) | 3 years
Target Vessel Revascularization (TVR) | ≤ 7 days post index procedure (In-hospital )
  TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion which includes upstream and downstream branches and the target lesion itself.
Target Vessel Revascularization (TVR) | 30 days
Target Vessel Revascularization (TVR) | 180 days
Target Vessel Revascularization (TVR) | 1 year
Target Vessel Revascularization (TVR) | 2 years
Target Vessel Revascularization (TVR) | 3 years
All coronary revascularization | ≤ 7 days post index procedure (In-hospital )
All coronary revascularization | 30 days
All coronary revascularization | 180 days
All coronary revascularization | 1 year
All coronary revascularization | 2 years
All coronary revascularization | 3 years
Scaffold thrombosis (per ARC definition) | Acute (0 - 24 hours post stent implantation) (Definite and Probable)
  Scaffold/Stent thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the catheterization lab.
  Timings:
  Acute scaffold/stent thrombosis : 0 - 24 hours post stent implantation Subacute scaffold/stent thrombosis: >24 hours - 30 days post stent implantation Late scaffold/stent thrombosis: 30 days - 1 year post stent implantation Very late scaffold/stent thrombosis: >1 year post stent implantation
Scaffold thrombosis (per ARC definition) | Subacute (>24 hours - 30 days post stent implantation)(Definite and Probable)
Scaffold thrombosis (per ARC definition) | Late (30 days - 1 year post stent implantation) (Definite and Probable)
Scaffold thrombosis (per ARC definition) | Very late (>1 year post stent implantation) (Definite and Probable)
Death/All Myocardial Infarction (MI) | ≤ 7 days post index procedure (In-hospital )
  All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in patients with coexisting potentially fatal non-cardiac disease (e.g. cancer, infection) should be classified as cardiac.
Death/All Myocardial Infarction (MI) | 30 days
Death/All Myocardial Infarction (MI) | 180 days
Death/All Myocardial Infarction (MI) | 1 year
Death/All Myocardial Infarction (MI) | 2 years
Death/All Myocardial Infarction (MI) | 3 years
Cardiac Death/All Myocardial Infarction (MI) | ≤ 7 days post index procedure (In-hospital )
  Cardiac death (CD): Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
Cardiac Death/All Myocardial Infarction (MI) | 30 days
Cardiac Death/All Myocardial Infarction (MI) | 180 days
Cardiac Death/All Myocardial Infarction (MI) | 1 year
Cardiac Death/All Myocardial Infarction (MI) | 2 years
Cardiac Death/All Myocardial Infarction (MI) | 3 years
Cardiac Death/All Myocardial Infarction (MI)/Target vessel revascularization (TVR) [Target vessel failure;TVF] | ≤ 7 days post index procedure (In-hospital )
Cardiac Death/All Myocardial Infarction (MI)/Target vessel revascularization (TVR) [TVF] | 30 days
Cardiac Death/All Myocardial Infarction (MI)/Target vessel revascularization (TVR) [TVF] | 180 days
Cardiac Death/All Myocardial Infarction (MI)/Target vessel revascularization (TVR) [TVF] | 1 year
Cardiac Death/All Myocardial Infarction (MI)/Target vessel revascularization (TVR) [TVF] | 2 years
Cardiac Death/All Myocardial Infarction (MI)/Target vessel revascularization (TVR) [TVF] | 3 years
Cardiac Death/TV MI/ID-TLR (Target lesion failure;TLF) | ≤ 7 days post index procedure (In-hospital )
Cardiac Death/TV MI/ID-TLR (TLF) | 30 days
Cardiac Death/TV MI/ID-TLR (TLF) | 180 days
Cardiac Death/TV MI/ID-TLR (TLF) | 1 year
Cardiac Death/TV MI/ID-TLR (TLF) | 2 years
Cardiac Death/TV MI/ID-TLR (TLF) | 3 years
Death/All Myocardial Infarction (MI)/All revascularization | ≤ 7 days post index procedure (In-hospital )
Death/All Myocardial Infarction (MI)/All revascularization | 30 days
Death/All Myocardial Infarction (MI)/All revascularization | 180 days
Death/All Myocardial Infarction (MI)/All revascularization | 1 year
Death/All Myocardial Infarction (MI)/All revascularization | 2 years
Death/All Myocardial Infarction (MI)/All revascularization | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Staehr, Study Director — Abbott Medical Devices
Locations (5):
- United States (5):
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Baptist Health Louisville, Louisville, Kentucky
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Turkey Creek Medical Center, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No